CLINICAL TRIAL: NCT05533775
Title: A Phase I/II, Open-Label, Single-Arm, Two-Part Trial to Evaluate Safety, Tolerability, Pharmacokinetics, and Anti-Tumor Activity of Glofitamab in Monotherapy and in Combination With Chemoimmunotherapy in Pediatric and Young Adult Participants With Relapsed/Refractory Mature B-Cell Non-Hodgkin Lymphoma
Brief Title: A Study to Evaluate Glofitamab Monotherapy and Glofitamab + Chemoimmunotherapy in Pediatric and Young Adult Participants With Relapsed/Refractory Mature B-Cell Non-Hodgkin Lymphoma
Acronym: iMATRIX GLO
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO43810
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Mature B-Cell Non-Hodgkin Lymphoma
Keywords: Relapsed; Refractory; Pediatrics; B-NHL
MeSH Terms: conditions — Recurrence | interventions — obinutuzumab; glofitamab; Rituximab; Ifosfamide; Carboplatin; Etoposide; tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Participants will receive glofitamab + R-ICE chemoimmunotherapy for up to 3 cycles (cycle length = 21 days).
  Interventions: Drug: Obinutuzumab; Drug: Glofitamab; Drug: Rituximab; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide; Drug: Tocilizumab
- Arm B (Experimental): Participants will receive glofitamab monotherapy for up to 12 cycles (cycle length = 21 days).
  Interventions: Drug: Obinutuzumab; Drug: Glofitamab; Drug: Tocilizumab

INTERVENTIONS:
Drug: Obinutuzumab — Participants will receive intravenous (IV) obinutuzumab pretreatment on Days 1 and 2 of Cycle 1 (Cycle length = 21 days)
Drug: Glofitamab — Arm A: Participants will receive IV glofitamab on Days 8 and 15 of Cycle 1, then on Day 1 of Cycles 2 and 3
  Arm B: Participants will receive IV glofitamab on Days 8 and 15 of Cycle 1, then on Day 1 of each cycle thereafter
  (Cycle length = 21 days)
Drug: Rituximab — Participants will receive IV rituximab on Days 5, 6, 7, and 8 of Cycles 2 and 3 (Cycle length = 21 days)
  Arms: Arm A
Drug: Ifosfamide — Participants will receive IV ifosfamide on Days 3, 4, and 5 of cycle 1 and on Days 5, 6, 7, and 8 of Cycles 2 and 3 (Cycle length = 21 days)
  Arms: Arm A
Drug: Carboplatin — Participants will receive IV carboplatin on Days 3, 4, and 5 of cycle 1 and on Days 5, 6, 7, and 8 of Cycles 2 and 3 (Cycle length = 21 days)
  Arms: Arm A
Drug: Etoposide — Participants will receive IV etoposide on Days 3, 4, and 5 of cycle 1 and on Days 5, 6, 7, and 8 of Cycles 2 and 3 (Cycle length = 21 days)
  Arms: Arm A
Drug: Tocilizumab — Participants will receive IV tocilizumab as needed to manage cytokine release syndrome (CRS) events

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of glofitamab, as monotherapy and in combination with a standard chemoimmunotherapy regimen: rituximab, ifosfamide, carboplatin, and etoposide (R-ICE) in pediatric and young adult participants with relapsed and refractory (R/R) mature B-cell non-Hodgkin lymphoma (B-NHL).

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to < 18 years at the time of signing Informed Consent for Cohort A Part 1 and Cohort B of the study, and age 6 months to < 30 years old at the time of signing Informed Consent for Cohort A Part 2 of the study
* Histologically re-confirmed diagnosis, via tissue biopsy, or bone marrow aspirate, pleural effusion, or ascites, prior to study entry of aggressive mature B-NHL that expresses CD20 (reconfirmed by IHC or flow cytometry if IHC is not possible), including BL, BAL (mature B-cell leukemia FAB L3), DLBCL, and PMBCL, at the time of first R/R disease for Cohort A and second or greater R/R disease for Cohort B
* Refractory or relapsed disease (i.e., prior treatment was ineffective or intolerable) following first-line standard-of-care chemoimmunotherapy for Cohort A and following at least two prior systemic chemoimmunotherapy regimens and who have exhausted all available established therapies for Cohort B
* Measurable disease, defined as: At least one bi-dimensionally measurable nodal lesion, defined as > 1.5 cm in its longest dimension, or at least one bi dimensionally measurable extranodal lesion, defined as > 1.0 cm in its longest dimension; or percentage of bone marrow involvement with lymphoma cells defined by cytomorphological analysis of bone marrow aspirates
* Adequate performance status, as assessed according to the Lansky or Karnofsky Performance Status scales: Participants < 16 years old: Lansky Performance Status ≥ 50%; Participants ≥ 16 years old: Karnofsky Performance Status ≥ 50%
* Adequate bone marrow, liver, and renal function
* Negative test results for acute or chronic hepatitis B virus (HBV), hepatitis C virus (HCV)
* Negative HIV test at screening, with the following exception: Individuals with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy for at least 4 weeks, have a CD4 count ≥200/uL, have an undetectable viral load, and have not had a history of opportunistic infection attributable to AIDS within the last 12 months
* Negative SARS-CoV-2 antigen or PCR test within 7 days prior to enrollment
* Participants and/or caregivers who are willing and able to complete clinical outcome assessments throughout the study using either paper or interviewer methods

Exclusion Criteria:

* Isolated CNS disease of mature B-NHL without systemic involvement, and primary CNS lymphoma
* Receipt of glofitamab prior to study enrollment
* Ongoing adverse events from prior anti-cancer therapy that were not resolved to Grade ≤ 1 (exceptions: alopecia, Grade 2 peripheral neuropathy)
* Grade ≥ 3 adverse events, with the exception of Grade 3 endocrinopathy managed with replacement therapy
* Participants with active infections which are not resolved prior to Day 1 of Cycle 1
* Prior solid organ transplantation
* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH), or chronic active Epstein-Barr viral infection (CAEBV)
* Active autoimmune disease requiring treatment
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (or recombinant antibody-related fusion proteins) or known sensitivity or allergy to murine products, except if the participant was able to safely receive it after initial administration (consider consultation with Medical Monitor)
* History of confirmed progressive multifocal leukoencephalopathy
* Current or past history of uncontrolled non-malignant CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease
* Evidence of significant and uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results
* Major surgery or significant traumatic injury < 28 days prior to the obinutuzumab pretreatment infusion (excluding biopsies) or anticipation of the need for major surgery during study treatment
* Administration of a live, attenuated vaccine within 4 weeks before the start of study treatment (obinutuzumab pretreatment) or at any time during the study treatment period and within 12 months after end of study treatment
* Participants with any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug

Ages: 6 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2032-11-30 (Estimated)

PRIMARY OUTCOMES:
Achievement of a complete response (CR) as determined by the investigator according to the International Pediatric NHL Response Criteria for pediatric participants and Lugano Classification for young adult participants (Arm A) | Up to 3 treatment cycles (cycle length = 21 days)
Percentage of participants with adverse events (AEs) (Arm A) | Approximately 3 years
Serum concentration of glofitamab in combination with R-ICE chemoimmunotherapy (Arm A) | Up to 3 treatment cycles (cycle length = 21 days)
Serum concentration of glofitamab monotherapy (Arm B) | Up to 12 treatment cycles (Arm B) (cycle length = 21 days)

SECONDARY OUTCOMES:
Objective response rate (ORR) (Arms A and B) | Up to 3 (Arm A) or 12 (Arm B) treatment cycles (cycle length = 21 days)
Duration of complete response (DOCR) (Arm A) | From the first occurrence of a documented complete response (CR) to documented disease progression or death from any cause (whichever occurs first) (approximately 3 years)
Progression-free survival (PFS) (Arm A) | From enrollment to the first occurrence of disease progression or death from any cause (whichever occurs first) (approximately 3 years)
Event-free survival (EFS) (Arm A) | From enrollment to the first occurrence of disease progression, death from any cause, or start of new anti-lymphoma therapy (not including planned hematopoietic stem cell transplantation (HSCT)) (approximately 3 years)
Overall survival (OS) (Arms A and B) | From enrollment to the date of death from any cause (Arm A = approximately 3 years, Arm B = approximately 4 years)
Percentage of participants who proceed to HSCT after up to three cycles of treatment (Arm A) | Up to 3 treatment cycles (cycle length = 21 days)
Duration of response (DOR) (Arm B) | From the first occurrence of a documented CR or partial response (PR) until documented disease progression or death from any cause, whichever occurs first (approximately 4 years)
Percentage of participants with AEs (arm B) | Approximately 3 years
Serum concentration of obinutuzumab (Arms A and B) | Up to 3 (Arm A) or 12 (Arm B) treatment cycles (cycle length = 21 days)
Serum concentration of rituximab (Arm A) | Up to 3 treatment cycles (cycle length = 21 days)
Percentage of participants with anti-drug antibodies (ADAs) (Arms A and B) | Up to 3 treatment cycles (cycle length = 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-LaRoche
Locations (28):
- United States (10):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente Oakland Medical Center, Oakland, California
  - Kaiser Permanente - Roseville, Roseville, California
  - Kaiser Permanente - Santa Clara, Santa Clara, California
  - Johns Hopkins University, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Childrens Mercy Hosp & Clinics, Kansas City, Missouri
  - MSKCC, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
- Australia (2):
  - Queensland Children?s Hospital, South Brisbane, Queensland
  - Perth Children's Hospital, Nedlands, Western Australia
- Brazil (2):
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Graacc-Grupo de Apoio ao adolescente e a crianca com cancer, São Paulo, São Paulo
- Sun Yet-sen University Cancer Center, Guangzhou, China
- Fakultni nemocnice v Motole;Klinika detske hematologie a onkologie, Prague, Czechia
- Rigshospitalet, København Ø, Denmark
- France (2):
  - Hôpital Pellegrin, Bordeaux
  - Gustave Roussy, Villejuif
- Universitaetsklinikum Muenster, Münster, Germany
- Semmelweis Egyetem II. sz. Gyermekgyogyaszati Klinika, Budapest, Hungary
- Italy (2):
  - IRCCS Ospedale Pediatrico Bambino Gesù, Rome, Lazio
  - Ospedaliera Ospedale Infantile Regina Margherita, Turin, Piedmont
- Ponadregionalne Centrum Onkologii Dzieci?cej ,,Przyladek Nadziei?;Klinika Transplantacji Szpiku, Onkologii i Hematologii Dzieciecej we Wroclawiu, Wroclaw, Poland
- South Korea (2):
  - Seoul National University Hospital- Pediatric Site, Seoul
  - Asan Medical Center, Seoul
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Infantil Universitario Niño Jesus, Madrid

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing